CLINICAL TRIAL: NCT01601626
Title: A Randomized, Phase 2b Study of a Double-Dose Lopinavir/Ritonavir-Based Antiretroviral Regimen With Rifampin-Based Tuberculosis Treatment Versus a Standard-Dose Lopinavir/Ritonavir-Based Antiretroviral Regimen With Rifabutin-Based Tuberculosis Treatment With or Without Raltegravir in HIV-1-Infected Persons Requiring Treatment for Active TB and HIV
Brief Title: Rifampin-Based Tuberculosis Treatment Versus Rifabutin-Based Tuberculosis Treatment in Persons With HIV
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped early due to feasibility concerns.
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5290; 1U01AI068636 (NIH)
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: HIV Infection; Tuberculosis
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Lopinavir; Ritonavir; lopinavir-ritonavir drug combination; Raltegravir Potassium; Isoniazid; Pyridoxine; Vitamin B 6; Pyrazinamide; Ethambutol; Rifabutin; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A: Standard-dose LPV/r w/RBT (Experimental): ART: lopinavir 400 mg/ritonavir 100 mg twice daily + two nucleoside reverse transcriptase inhibitors.
  Anti-TB therapy: isoniazid 300 mg, rifabutin 300 mg, weight-based dosing for ethambutol and pyrazinamide, and pyridoxine 25 mg daily.
  After completion of TB treatment through week 72: lopinavir 400 mg/ritonavir 100 mg twice daily + two nucleoside reverse transcriptase inhibitors (NRTIs).
  Interventions: Drug: Standard-dose Lopinavir/Ritonavir; Drug: Isoniazid; Drug: Pyridoxine; Drug: Pyrazinamide; Drug: Ethambutol; Drug: Rifabutin
- B: Double-dose LPV/r w/RIF (Active Comparator): ART: lopinavir 800 mg/ritonavir 200 mg twice daily + two nucleoside reverse transcriptase inhibitors.
  Anti-TB therapy: isoniazid 300 mg, weight-based dosing for rifampin, ethambutol, and pyrazinamide, and pyridoxine 25 mg daily.
  After completion of TB treatment through week 72: lopinavir 400 mg/ritonavir 100 mg twice daily + two nucleoside reverse transcriptase inhibitors (NRTIs).
  Interventions: Drug: Double-dose Lopinavir/Ritonavir; Drug: Isoniazid; Drug: Pyridoxine; Drug: Pyrazinamide; Drug: Ethambutol; Drug: Rifampin
- C: Standard-Dose LPV/r w/RBT + RAL (Experimental): ART: lopinavir 400 mg/ritonavir 100 mg twice daily + raltegravir 400 mg twice daily + two nucleoside reverse transcriptase inhibitors.
  Anti-TB therapy: isoniazid 300 mg, rifabutin 300 mg, weight-based dosing for ethambutol and pyrazinamide, and pyridoxine 25 mg daily.
  After completion of TB treatment through week 72: lopinavir 400 mg/ritonavir 100 mg twice daily + two nucleoside reverse transcriptase inhibitors (NRTIs).
  Interventions: Drug: Standard-dose Lopinavir/Ritonavir; Drug: Raltegravir; Drug: Isoniazid; Drug: Pyridoxine; Drug: Pyrazinamide; Drug: Ethambutol; Drug: Rifabutin

INTERVENTIONS:
Drug: Standard-dose Lopinavir/Ritonavir — Two LPV 200 mg/RTV 50 mg fixed-dose combination tablets orally twice daily from entry to Week 72.
  Other Names: LPV/RTV; LPV/r; Aluvia; Kaletra
  Arms: A: Standard-dose LPV/r w/RBT; C: Standard-Dose LPV/r w/RBT + RAL
Drug: Double-dose Lopinavir/Ritonavir — Four LPV 200 mg/RTV 50 mg fixed-dose combination tablets orally twice daily from entry through Week 72.
  Other Names: LPV/RTV; LPV/r; Aluvia; Kaletra
  Arms: B: Double-dose LPV/r w/RIF
Drug: Raltegravir — One 400 mg tablet orally twice daily from entry to Week 72.
  Other Names: RAL; Isentress
  Arms: C: Standard-Dose LPV/r w/RBT + RAL
Drug: Isoniazid — 300 mg orally once daily from entry through Week 24.
  Other Names: INH
Drug: Pyridoxine — 25 mg orally once daily from entry to Week 24.
  Other Names: Vitamin B6
Drug: Pyrazinamide — 20 to 30 mg/kg orally once daily (not to exceed 2 g per day) from entry through Week 8 study visit (or until completion of intensive TB treatment as determined after dose adjustment in accrual period 1 participants).
  Other Names: PZA
Drug: Ethambutol — 15 to 20 mg/kg orally once daily from entry through Week 8 study visit (or until completion of intensive TB treatment as determined after dose adjustment in accrual period 1 participants).
  Other Names: EMB
Drug: Rifabutin — 300 mg of rifabutin orally once until LPV/RTV is started; then the dose will be reduced to 150 mg daily from the start of LPV/RTV through Week 24.
  Other Names: RBT
  Arms: A: Standard-dose LPV/r w/RBT; C: Standard-Dose LPV/r w/RBT + RAL
Drug: Rifampin — Weight-based dose; for weight < 45 kg: 450 mg orally once daily; for weight > 45 kg: 600 mg orally once daily, from entry to week 24.
  Other Names: RIF
  Arms: B: Double-dose LPV/r w/RIF

SUMMARY:
There is a rapidly-growing need to identify evidence-based, safe, and effective co-treatment regimens for HIV-related tuberculosis (TB) among patients who require protease inhibitor (PI)-based antiretroviral therapy (ART). This study compared three alternative co-treatment options among participants in high TB endemic resource-constrained settings, in which one co-treatment option explores if an additional anti-HIV drug needs to be used when patients are being treated with a PI together with rifabutin-based anti-TB treatment.

DETAILED DESCRIPTION:
Rifampin (RIF), the cornerstone of TB treatment, has very problematic drug-drug interactions with PIs. The use of relatively high doses of ritonavir appear necessary to overcome this interaction, but it is unclear whether the co-treatment regimen of RIF-based TB treatment and double-dose PI-based ART will be safe and tolerable for patients with HIV-related TB and effective in treating both HIV and TB. The study proposed to determine if, for HIV-1-infected participants with active TB who require PI-based ART, a standard-dose lopinavir/ritonavir (LPV/r) regimen, with or without raltegravir (RAL), coupled with rifabutin (RBT)-based TB treatment is superior to a double-dose LPV/r regimen coupled with RIF-based TB treatment.

At study entry, participants were randomized (1:1:1) to receive standard-dose LPV/r-based HIV treatment plus RBT-based TB treatment (Arm A), double-dose LPV/r-based HIV treatment plus RIF-based TB treatment (Arm B), or standard-dose LPV/r-based HIV treatment plus RAL plus RBT-based TB treatment (Arm C).

Accrual was planned to take place in two accrual periods. Accrual period 1 would enroll 60 participants who would undergo an initial dose-finding period before continuing regular study follow-up. Once the review of the dose-finding pharmacokinetic (PK) and safety data from accrual period 1 participants was completed, accrual period 2 was planned to open to accrual.

Study duration was 72 weeks. Visits occurred at weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 72. The key evaluations included physical examination, clinical assessments, TB evaluations including chest x-ray, acid-fast bacilli (AFB) smear, mycobacterial culture, and drug susceptibility testing, CD4 cell count, HIV viral load, hematology, chemistry, and pregnancy testing in women of reproductive potential. Sputum, serum, and urine were stored for use in future analyses. An intensive PK visit occurred at day 12. PK blood draws in participants in Arms A and C were at RBT pre-dose and at 2, 4, 5, 6, and 24 hours RBT post-dose. PK blood draws in participants in Arm B were at LPV/r pre-dose and at 2, 4, 5, and 6 hours LPV/r post-dose.

The target sample size was 471 participants, but the study was terminated after 71 participants due to feasibility concerns. The 71 participants were followed for the planned 72 weeks. Because of the limited sample size, formal statistical comparisons were not undertaken as originally planned.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* CD4+/CD8+ T-cell count obtained within 30 days prior to study entry
* Confirmed or probable pulmonary or extrapulmonary TB (more information on the criterion can be found in the protocol)
* Chest x-ray within 30 days prior to study entry
* A PI-based antiretroviral regimen is required, as determined by the participant's primary clinician/clinical facility
* Certain laboratory values obtained within 14 days prior to study entry (more information on the criterion can be found in the protocol)
* For females of reproductive potential, negative serum or urine pregnancy test within 7 days prior to study entry and 72 hours of starting study medications
* Willing to use acceptable methods of contraception while on study drugs and for 6 weeks after stopping these drugs
* Karnofsky performance score > 40 within 14 days prior to study entry, and likelihood of survival, in the opinion of the site investigator, for at least 6 months
* Ability to swallow oral medications
* Ability and willingness of participant or legal guardian/representative to provide informed consent

Exclusion Criteria:

* History of completed TB treatment and resolution of TB symptoms less than 1 year prior to the current TB episode at study entry, or incomplete treatment for a prior episode of TB (i.e., defaulted past TB treatment) at any time prior to the current TB episode
* Documented multidrug-resistant tuberculosis (MDR TB) or extensively drug-resistant tuberculosis (XDR TB)
* Participants infected with a rifamycin resistant strain of TB (more information on the criterion can be found in the protocol)
* Receipt of more than 28 cumulative days of anti-TB treatment for the current TB episode prior to study entry
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Active illness requiring systemic treatment and/or hospitalization within 30 days prior to study entry, or that in the opinion of the site investigator, might otherwise interfere with adherence to study requirements
* Pregnant or breastfeeding
* Anticipated receipt of prohibited medications (more information on the criterion can be found in the protocol)
* Known intolerance/allergy/sensitivity or any hypersensitivity to components of study drugs or their formulations
* History of close contact with known MDR or XDR TB patients at any time prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-07-13 (Actual); Primary Completion 2017-01-19 (Actual); Study Completion 2017-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constance A Benson, MD, Study Chair — University of California, San Diego; Umesh Lalloo, MD, FRCP, Study Chair — Nelson R. Mandela School of Medicine
Locations (9):
- Brazil (2):
  - Hospital Nossa Senhora da Conceicao CRS (12201), Porto Alegre, Rio Grande do Sul
  - Instituto de Pesquisa Clinica Evandro Chagas (12101), Rio de Janeiro
- Haiti (2):
  - Les Centres GHESKIO CRS (30022), Port-au-Prince
  - GHESKIO Institute of Infectious Diseases and Reproductive Health (GHESKIO - IMIS) CRS (31730), Port-au-Prince
- Moi University Clinical Research Center CRS (12601), Eldoret, Kenya
- Peru (2):
  - Investigaciones Medicas en Salud (INMENSA) (11302), San Isidro, Lima region
  - Asociacion Civil Impacta Salud y Educacion - Miraf CRS (11301), Lima
- South Africa (2):
  - Wits HIV CRS (11101), Johannesburg, Gauteng
  - Durban Adult HIV CRS (11201), Durban

REFERENCES:
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004; Clarification, August 2009 — https://rsc.tech-res.com/docs/default-source/safety/table_for_grading_severity_of_adult_pediatric_adverse_events.pdf
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.tech-res.com/docs/default-source/safety/manual_for_expedited_reporting_aes_to_daids_v2.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited at 9 sites from 5 countries (2 each from Brazil, Haiti, Peru, and South Africa and 1 from Kenya) between July 2013 and February 2016.
Groups:
- A: Standard-dose LPV/r w/RBT: ART: standard-dose LPV/r twice daily + two NRTIs. Anti-TB therapy: isoniazid, rifabutin, ethambutol, pyrazinamide, and pyridoxine daily.
  After completion of TB treatment through week 72: standard-dose LPV/r twice daily + two NRTIs.
- B: Double-dose LPV/r w/RIF: ART: double-dose LPV/r twice daily + 2 NRTIs. Anti-TB therapy: isoniazid, rifampin, ethambutol, pyrazinamide, and pyridoxine daily.
  After completion of TB treatment through week 72: standard-dose LPV/r twice daily + 2 NRTIs.
- C: Standard-Dose LPV/r + RAL w/RBT: ART: standard-dose LPV/r twice daily + RAL + two NRTIs. Anti-TB therapy: isoniazid, rifabutin, ethambutol, pyrazinamide, and pyridoxine daily.
  After completion of TB treatment through week 72: standard-dose LPV/r twice daily + RAL + two NRTIs.
Period: Overall Study
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Started | 24 | 24 | 23
Completed | 21 | 19 | 21
Not Completed | 3 | 5 | 2
Not completed — Death | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Unable to Get to Clinic | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Not Willing to Adhere to Requirements | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants were included.
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT | Total
Number analyzed (Participants) | 24 | 24 | 23 | 71
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 42 [33 to 49] | 35 [29 to 41] | 38 [32 to 47] | 37 [32 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 15 | 37
  Male | 11 | 15 | 8 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black of African Origin | 7 | 8 | 6 | 21
  Black African | 8 | 6 | 4 | 18
  White | 4 | 2 | 6 | 12
  Mixed Black | 3 | 5 | 3 | 11
  Mestizo | 2 | 2 | 2 | 6
  Mixed, of Predominantly African Ancestry | 0 | 0 | 1 | 1
  Other | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Haiti | 6 | 6 | 6 | 18
  Brazil | 8 | 10 | 10 | 28
  South Africa | 4 | 3 | 3 | 10
  Kenya | 4 | 3 | 2 | 9
  Peru | 2 | 2 | 2 | 6
Qualitative HIV RNA [Count of Participants; unit: Participants] — The lower limit of quantification of the HIV RNA assay used in the protocol was 40 copies/mL.
  Participants
    Less than 40 copies/mL | 4 | 2 | 3 | 9
    Greater than or equal to 40 copies/mL | 20 | 22 | 20 | 62
Quantitative HIV RNA [Median (Inter-Quartile Range); unit: log10 copies/mL] — The lower limit of quantification of the HIV RNA assay used in the protocol was 40 copies/mL. Population: Quantitative HIV RNA was summarized in the participants whose HIV RNA was above the assay's lower limit of quantification.
  log10 copies/mL
    number analyzed (Participants) | 20 | 22 | 20 | 62
    (all) | 4.7 [3.4 to 5.6] | 4.8 [4.2 to 5.3] | 4.2 [3.2 to 5.0] | 4.6 [3.5 to 5.3]
CD4 Cell Count [Median (Inter-Quartile Range); unit: cells/mm^3] | 128 [60 to 234] | 117 [51 to 246] | 158 [73 to 202] | 130 [55 to 231]
Tuberculosis (TB) Diagnosis Certainty [Count of Participants; unit: Participants] — The protocol document contains the definitions of confirmed and probable for pulmonary and extrapulmonary TB in section 4.1.3.
  Participants
    Confirmed Pulmonary TB | 13 | 8 | 6 | 27
    Confirmed Extrapulmonary TB | 1 | 1 | 3 | 5
    Confirmed Pulmonary and Extrapulmonary TB | 1 | 0 | 0 | 1
    Probable Pulmonary TB | 9 | 15 | 13 | 37
    Probable Extrapulmonary TB | 0 | 0 | 1 | 1
Acid Fast Bacilli (AFB) Smear [Count of Participants; unit: Participants]
  Positive | 11 | 8 | 6 | 25
  Negative | 10 | 14 | 16 | 40
  No Results Available | 3 | 2 | 1 | 6
Mycobacteria Tuberculosis (MTB) Culture [Count of Participants; unit: Participants]
  MTB-Positive | 13 | 8 | 9 | 30
  MTB-Negative | 6 | 13 | 13 | 32
  No Results Available | 5 | 3 | 1 | 9
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 19.9 [18.3 to 22.1] | 20.4 [17.9 to 21.5] | 18.9 [17.9 to 21.5] | 19.6 [17.9 to 21.5]

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Whose HIV Viral Load Was Less Than 400 Copies/mL at Week 48.
Description: The percent of participants whose HIV viral load was less than 400 copies/mL at week 48 was calculated with an associated standard error. The confidence interval was calculated using Wilson's score method. Participants who were lost-to-follow-up or dead by week 48 or had missing results at week 48 were coded as having HIV viral load greater than 400 copies/mL. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: 48 weeks
Population: All randomized participants were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 24 | 24 | 23
percentage of participants | 58.3 [38.8 to 75.5] | 66.7 [46.7 to 82.0] | 60.9 [40.8 to 77.8]

2. Secondary Outcome: Percent of Participants Who Experienced Sputum Conversion at Week 8.
Description: Sputum conversion was defined as culture MTB-negative at week 8 or AFB smear negative at week 8 (and culture contaminated or missing at week 8); there were no Xpert MTB/RIF results at week 8. The percent of participants experienced sputum conversion at week 8 was calculated with an associated standard error. The confidence interval was calculated using Wilson's score method. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: 8 weeks
Population: Participants who were either culture MTB-positive at entry; AFB smear positive at entry (and culture MTB-negative, contaminated, or missing at entry); or Xpert MTB/RIF positive at entry (and culture or smear negative, contaminated, or missing at entry) were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 16 | 11 | 10
percentage of participants | 87.5 [64.0 to 96.5] | 81.8 [52.3 to 94.9] | 70.0 [39.7 to 89.2]

3. Secondary Outcome: Percent of Participants Who Experienced TB Treatment Failure
Description: TB treatment failure was defined as having a MTB-positive culture after 16 weeks of TB treatment for a participant who was documented to be taking TB medications. The percent of participants who experienced TB treatment failure was calculated with an associated standard error. The confidence interval was calculated using Wilson's score method. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: After 16 weeks and through week 72
Population: All randomized participants were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 24 | 24 | 23
percentage of participants | 0.0 [0.0 to 13.8] | 0.0 [0.0 to 13.8] | 0.0 [0.0 to 14.3]

4. Secondary Outcome: Percent of Participants Who Experienced TB Relapse/Recurrence
Description: TB relapse/recurrence was defined as having had 2 consecutive MTB-negative cultures and subsequently had clinical or radiographic deterioration consistent with active TB at or after week 24 and before week 72. The percent of participants who experienced TB relapse/recurrence was calculated with an associated standard error. The confidence interval was calculated using Wilson's score method. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: At or after 24 weeks and through week 72
Population: All randomized participants were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 24 | 24 | 23
percentage of participants | 0.0 [0.0 to 13.8] | 4.2 [0.7 to 20.2] | 4.3 [0.8 to 21.0]

5. Secondary Outcome: Percent of Participants Who Experienced TB Relapse/Recurrence and Who Had TB Drug Resistance
Description: TB relapse/recurrence was defined as having had 2 consecutive MTB-negative cultures and subsequently had clinical or radiographic deterioration consistent with active TB at or after week 24 and before week 72. The drug resistance was determined based on phenotypic methods. The percent of participants who experienced TB relapse/recurrence and who had TB drug resistance was calculated with an associated standard error. The confidence interval was calculated using Wilson's score method. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: At or after 24 weeks and through week 72
Population: All participants who experienced TB relapse/recurrence were included.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 0 | 1 | 1
participants |  | 0 [0.0 to 79.3] | 0 [0.0 to 32.4]

6. Secondary Outcome: Percent of Participants Whose HIV Viral Load Was Less Than 50 Copies/mL at Week 48
Description: The percent of participants whose HIV viral load was less than 50 copies/mL at week 48 was calculated with an associated standard error. Participants who were lost-to-follow-up or dead by week 48 or had missing RNA at week 48 were coded as having HIV viral load greater than 50 copies/mL. The confidence interval was calculated using Wilson's score method. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: 48 weeks
Population: All randomized participants were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 24 | 24 | 23
percentage of participants | 45.8 [27.9 to 64.9] | 54.2 [35.1 to 72.1] | 56.5 [36.8 to 74.4]

7. Secondary Outcome: Number of Participants Reporting a Grade 3 or 4 Sign or Symptom
Description: The number of participants reporting a grade 3 (severe) or grade 4 (life-threatening) sign or symptom were summarized. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: After randomization and through week 72
Population: All randomized participants were included.
Measure: Count of Participants; unit: Participants
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 24 | 24 | 23
Participants | 7 | 5 | 5

8. Secondary Outcome: Number of Participants Reporting a Grade 3 or 4 Laboratory Abnormality
Description: The number of participants reporting a grade 3 (severe) or grade 4 (life-threatening) laboratory abnormality were summarized. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: After randomization and through week 72
Population: All randomized participants were included.
Measure: Count of Participants; unit: Participants
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 24 | 24 | 23
Participants | 6 | 3 | 5

9. Secondary Outcome: Percent of Participants Who Interrupted or Discontinued at Least One HIV Drug Due to Toxicity
Description: The percent of participants who interrupted or discontinued at least one HIV drug due to toxicity was calculated with an associated standard error. The confidence interval was calculated using Wilson's score method. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: After randomization and through week 72
Population: All randomized participants were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 24 | 24 | 23
percentage of participants | 20.8 [9.2 to 40.5] | 16.7 [6.7 to 35.9] | 21.7 [9.7 to 41.9]

10. Secondary Outcome: Percent of Participants Who Interrupted or Discontinued at Least One TB Drug Due to Toxicity
Description: The percent of participants who interrupted or discontinued at least one TB drug due to toxicity was calculated with an associated standard error. The confidence interval was calculated using Wilson's score method. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: After randomization and through to the discontinuation of the last TB drug
Population: All randomized participants were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 24 | 24 | 23
percentage of participants | 20.8 [9.2 to 40.5] | 8.3 [2.3 to 25.8] | 13.0 [4.5 to 32.1]

11. Secondary Outcome: Percent of Participants Who Experienced HIV Virologic Failure
Description: Virologic failure was defined as the occurrence of two consecutive plasma HIV-1 RNA levels ≥1000 copies/mL at or after 16 weeks and within 24 weeks of treatment initiation or ≥400 copies/mL at or after 24 weeks of treatment, regardless of whether randomized ART was being taken at the time of virologic failure. Participants who were missing data due to being lost-to-follow-up or dead were coded as virologic failures. The percent of participants who experienced HIV virologic failure was calculated with an associated standard error. The confidence interval was calculated using Wilson's score method. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: At weeks 16, 24, 48, and 72
Population: All randomized participants were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 24 | 24 | 23
percentage of participants | 29.2 [14.9 to 49.2] | 50.0 [31.4 to 68.6] | 30.4 [15.6 to 50.9]

12. Secondary Outcome: Cumulative Probability of HIV Virologic Failure at Week 72
Description: Virologic failure was defined as the occurrence of two consecutive plasma HIV-1 RNA levels ≥1000 copies/mL at or after 16 weeks and within 24 weeks of treatment initiation or ≥400 copies/mL at or after 24 weeks of treatment, regardless of whether randomized ART was being taken at the time of virologic failure. The percent of participants with HIV virologic failure at week 72 was calculated using a Kaplan-Meier estimator with an associated standard error. The confidence interval was calculated using a log-log transformation. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: At weeks 16, 24, 48, and 72
Population: All randomized participants were included.
Measure: Number (95% Confidence Interval); unit: cumulative events per 100 participants
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 24 | 24 | 23
cumulative events per 100 participants | 29.2 [15.1 to 51.6] | 50.0 [32.2 to 70.9] | 30.4 [15.8 to 53.4]

13. Secondary Outcome: Number of Participants Who Experienced MTB IRIS
Description: The number of participants who experienced MTB immune reconstitution inflammatory syndrome (IRIS) was summarized. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: After randomization and through week 72
Population: All randomized participants were included.
Measure: Count of Participants; unit: Participants
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 24 | 24 | 23
Participants | 1 | 2 | 3

14. Secondary Outcome: CD4 Count Change From Baseline to Week 8
Description: The difference in CD4 count from baseline to week 8 was calculated as the CD4 count at week 8 minus the CD4 count at baseline. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: Baseline and 8 weeks
Population: Participants who had CD4 cell count data available at baseline and week 8 were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 22 | 24 | 22
cells/mm^3 | 7 [-71 to 33] | 26 [2 to 106] | 37 [-60 to 79]

15. Secondary Outcome: CD4 Count Change From Baseline to Week 24
Description: The difference in CD4 count from baseline to week 24 was calculated as the CD4 count at week 24 minus the CD4 count at baseline. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: Baseline and 24 weeks
Population: Participants who had CD4 cell count data available at baseline and week 24 were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 21 | 23 | 18
cells/mm^3 | 20 [-38 to 56] | 56 [12 to 110] | 13 [-64 to 100]

16. Secondary Outcome: CD4 Count Change From Baseline to Week 48
Description: The difference in CD4 count from baseline to week 48 was calculated as the CD4 count at week 48 minus the CD4 count at baseline. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: Baseline and 48 weeks
Population: Participants who had CD4 cell count data available at baseline and week 48 were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 20 | 20 | 18
cells/mm^3 | 99 [1 to 159] | 119 [57 to 263] | 74 [16 to 115]

17. Secondary Outcome: CD4 Count Change From Baseline to Week 72
Description: The difference in CD4 count from baseline to week 72 was calculated as the CD4 count at week 72 minus the CD4 count at baseline. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: Baseline and 72 weeks
Population: Participants who had CD4 cell count data available at baseline and week 72 were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 20 | 19 | 20
cells/mm^3 | 126 [26 to 247] | 212 [93 to 281] | 54 [-6 to 203]

18. Secondary Outcome: Percent of Participants Who Experienced a New AIDS-defining Illness
Description: New post-randomization diagnoses were considered AIDS-defining based on the CDC classification system. The percent of participants who experienced a new AIDS-defining illness was calculated with an associated standard error. The confidence interval was calculated using Wilson's score method. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: After randomization and through week 72
Population: All randomized participants were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 24 | 24 | 23
percentage of participants | 0.0 [0.0 to 13.8] | 4.2 [0.7 to 20.2] | 0.0 [0.0 to 14.3]

19. Secondary Outcome: Percent of Participants Who Died
Description: The percent of participants who died was calculated with an associated standard error. Confidence intervals were calculated using Wilson's score method. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: After randomization and through week 72
Population: All randomized participants were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 24 | 24 | 23
percentage of participants | 4.2 [0.7 to 20.2] | 4.7 [0.7 to 20.2] | 4.3 [0.8 to 21.0]

20. Secondary Outcome: Percent of Participants Who Experienced a New AIDS-defining Illness or Died
Description: New post-randomization diagnoses were considered AIDS-defining based on the CDC classification system. The percent of participants who experienced a new AIDS-defining illness or died was calculated with an associated standard error. Confidence intervals were calculated using Wilson's score method. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: After randomization and through week 72
Population: All randomized participants were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 24 | 24 | 23
percentage of participants | 4.2 [0.7 to 20.2] | 8.3 [2.3 to 25.8] | 4.3 [0.8 to 21.0]

21. Other Pre Specified Outcome: LPV Cmax and Cmin in Participants Enrolled in Arms A, B, and C
Description: Describe LPV plasma pharmacokinetic (PK) characteristics (maximum concentration [Cmax] and minimum concentration [Cmin]) in participants enrolled in Arms A, B, and C, determined by non-compartmental analysis of 12-hour PK sampling. The pre-dose concentration was determined using a sample drawn 12 hours after the previous LPV dose and was used as the 12-hour LPV concentration. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: At 2 weeks: pre-dose and at 2, 4, 5, and 6 hours post-dose
Population: Participants were included in this analysis if they completed the PK visit, did not miss any doses of any study-required medications on the day prior to the PK visit, and the LPV concentration at the pre-dose draw was above the assay's lower limit of quantification (20 ng/mL).
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 19 | 17 | 14
ng/mL
  Maximum Concentration (Cmax) | 18531 [12978 to 21627] | 18138 [11366 to 22807] | 16802 [12609 to 24924]
  Minimum Concentration (Cmin) | 9920 [2421 to 16127] | 8033 [4061 to 9481] | 8548 [5603 to 15968]

22. Other Pre Specified Outcome: LPV AUC in Participants Enrolled in Arms A, B, and C
Description: Describe LPV plasma PK characteristics (area under the curve [AUC] between 0 and 12 hours) in participants enrolled in Arms A, B, and C, determined by non-compartmental analysis of 12-hour PK sampling. The pre-dose concentration was determined using a sample drawn 12 hours after the previous LPV dose and was used as the 12-hour LPV concentration. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: At 2 weeks: pre-dose and at 2, 4, 5, and 6 hours post-dose
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: hours*ng/mL
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 19 | 17 | 14
hours*ng/mL | 159796 [113493 to 222251] | 161772 [102118 to 209509] | 149247 [122324 to 243273]

23. Other Pre Specified Outcome: RBT Cmax and Cmin in Participants Enrolled in Arms A and C
Description: Describe RBT plasma PK characteristics (Cmax and Cmin) in participants enrolled in Arms A and C, determined by non-compartmental analysis of 24-hour PK sampling. The pre-dose concentration was determined using a sample drawn 24 hours after the previous RBT dose. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: At 2 weeks: pre-dose and at 2, 4, 5, 6, and 24 hours post-dose
Population: Participants were included in this analysis if they completed the PK visit, did not miss any doses of any study-required medications on the day prior to the PK visit, followed the protocol-required RBT dosing schedule, and the RBT concentration at the pre-dose draw was above the assay's lower limit of quantification (75 ng/mL).
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 18 | 0 | 11
ng/mL
  Maximum Concentration (Cmax) | 461 [361 to 625] |  | 349 [249 to 505]
  Minimum Concentration (Cmin) | 161 [104 to 255] |  | 115 [88 to 171]

24. Other Pre Specified Outcome: RBT AUC in Participants Enrolled in Arms A and C
Description: Describe RBT plasma PK characteristics (area under the curve [AUC] between 0 and 24 hours) in participants enrolled in Arms A and C, determined by non-compartmental analysis of 24-hour PK sampling. The pre-dose concentration was determined using a sample drawn 24 hours after the previous RBT dose. As stated in the Detailed Study Description of the Protocol Section, formal statistical comparisons were not undertaken because of limited sample size.
Time Frame: At 2 weeks: pre-dose and at 2, 4, 5, 6, and 24 hours post-dose
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: hours*ng/mL
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 18 | 0 | 11
hours*ng/mL | 7374 [5909 to 11785] |  | 5516 [4147 to 7060]

25. Other Pre Specified Outcome: RAL Cmax and Cmin in Participants Enrolled in Arm C
Description: Describe RAL plasma PK characteristics (Cmax and Cmin) in participants enrolled in Arm C, determined by non-compartmental analysis of 24-hour PK sampling. The pre-dose concentration was determined using a sample drawn 12 hours after the previous RAL dose and was used as the 12-hour RAL concentration.
Time Frame: At 2 weeks: pre-dose and at 2, 4, 5, 6, and 24 hours post-dose
Population: Participants were included in this analysis if they completed the PK visit, did not miss any doses of any study-required medications on the day prior to the PK visit, and the RAL concentration at the pre-dose draw was above the assay's lower limit of quantification (5 ng/mL).
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 0 | 0 | 16
ng/mL
  Maximum Concentration (Cmax) |  |  | 2830 [469 to 4560]
  Minimum Concentration (Cmin) |  |  | 166 [53 to 197]

26. Other Pre Specified Outcome: RAL AUC in Participants Enrolled in Arm C
Description: Describe RAL plasma PK characteristics (area under the curve [AUC] between 0 and 24 hours) in participants enrolled in Arm C, determined by non-compartmental analysis of 24-hour PK sampling. The pre-dose concentration was determined using a sample drawn 12 hours after the previous RAL dose and was used as the 12-hour RAL concentration.
Time Frame: At 2 weeks: pre-dose and at 2, 4, 5, 6, and 24 hours post-dose
Population: as for outcome 25
Measure: Median (Inter-Quartile Range); unit: hours*ng/mL
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
Number analyzed (Participants) | 0 | 0 | 16
hours*ng/mL |  |  | 11338 [2618 to 15363]

ADVERSE EVENTS:
Time Frame: From study entry to either premature study discontinuation or study completion at Week 72.
Description: The study protocol required reporting of all new diagnoses; all new Grade 2 (moderate) or higher TB-related signs and symptoms, all new signs and symptoms Grade 3 (severe) or higher; all new all Grade 3 or higher laboratory values; and all signs, symptoms, and laboratory values that led to a change in treatment, regardless of grade. The DAIDS AE Grading Table (V1.0) and EAE Manual (V2.0) were used. All randomized participants who initiated study treatment were included.
Arm/Group | A: Standard-dose LPV/r w/RBT | B: Double-dose LPV/r w/RIF | C: Standard-Dose LPV/r + RAL w/RBT
All-Cause Mortality (participants affected / at risk) | 1/24 | 1/24 | 1/23
Serious Adverse Events (participants affected / at risk) | 4/24 | 5/24 | 5/23
Other Adverse Events (participants affected / at risk) | 24/24 | 23/24 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: Standard-dose LPV/r w/RBT (N=24) | B: Double-dose LPV/r w/RIF (N=24) | C: Standard-Dose LPV/r + RAL w/RBT (N=23)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Iridocyclitis (Eye disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Acute hepatitis B (Infections and infestations) | 1 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Rhodococcus infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Tuberculosis gastrointestinal (Infections and infestations) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A: Standard-dose LPV/r w/RBT (N=24) | B: Double-dose LPV/r w/RIF (N=24) | C: Standard-Dose LPV/r + RAL w/RBT (N=23)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 2 | 2
Tachycardia (Cardiac disorders) | 1 | 2 | 3
Eye pain (Eye disorders) | 3 | 0 | 0
Ocular hyperaemia (Eye disorders) | 3 | 0 | 0
Uveitis (Eye disorders) | 2 | 0 | 0
Visual acuity reduced (Eye disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2
Oral disorder (Gastrointestinal disorders) | 3 | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2
Asthenia (General disorders) | 2 | 1 | 1
Chest pain (General disorders) | 2 | 1 | 1
Fatigue (General disorders) | 2 | 0 | 2
Pyrexia (General disorders) | 3 | 6 | 3
Immune reconstitution inflammatory syndrome associated tuberculosis (Infections and infestations) | 1 | 2 | 4
Oral candidiasis (Infections and infestations) | 3 | 3 | 2
Pneumonia bacterial (Infections and infestations) | 2 | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 2 | 0
Purulent discharge (Infections and infestations) | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 2 | 3 | 4
Aspartate aminotransferase increased (Investigations) | 7 | 7 | 9
Blood albumin decreased (Investigations) | 15 | 15 | 14
Blood alkaline phosphatase increased (Investigations) | 6 | 8 | 6
Blood bicarbonate decreased (Investigations) | 3 | 2 | 3
Blood bilirubin increased (Investigations) | 2 | 2 | 1
Blood creatinine increased (Investigations) | 3 | 1 | 1
Blood potassium decreased (Investigations) | 0 | 3 | 1
Blood potassium increased (Investigations) | 0 | 1 | 3
Blood sodium decreased (Investigations) | 8 | 8 | 11
Blood sodium increased (Investigations) | 3 | 5 | 4
Haemoglobin decreased (Investigations) | 14 | 9 | 7
Neutrophil count decreased (Investigations) | 3 | 1 | 3
Weight decreased (Investigations) | 2 | 3 | 3
White blood cell count decreased (Investigations) | 1 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Altered state of consciousness (Nervous system disorders) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 1
Headache (Nervous system disorders) | 2 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Blister (Skin and subcutaneous tissue disorders) | 1 | 2 | 1

LIMITATIONS AND CAVEATS:
The study was terminated after 71 of 471 participants enrolled. Therefore, the study was under-powered and formal statistical comparisons between study arms were not undertaken as originally planned. Instead, summaries within study arm were provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (3):
  • Statistical Analysis Plan: Primary Analysis (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT01601626/SAP_001.pdf
  • Statistical Analysis Plan: PK and Safety Interim Analysis (2016-10-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT01601626/SAP_002.pdf
  • Study Protocol and Informed Consent Form (2012-01-31): https://cdn.clinicaltrials.gov/large-docs/26/NCT01601626/Prot_ICF_003.pdf